CLINICAL TRIAL: NCT06278116
Title: Comparison of Absorbance Values, Sensory Evaluations and Periodontal Effects of Five Different Products for Clean Aligners Cleansing: Randomized Clinical Trial
Brief Title: Comparison of Absorbance Values, Sensory Evaluations and Periodontal Effects of Five Different Products for Clean Aligners Cleansing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Andrea Scribante, Associate Professor, Principal Investigator, University of Pavia
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2024-ALIGNERSCLEANSIGN
Record Dates: First submitted 2024-02-18; First posted 2024-02-26 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Dental Malocclusion
Keywords: clear aligners
MeSH Terms: conditions — Malocclusion | interventions — Water

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Water (Active Comparator)
  Interventions: Other: Aligners cleansing with water
- Dish soap (Active Comparator)
  Interventions: Other: Aligners cleansing with dish soap Svelto
- Polident Antibacterial Denture Cleaner® (Active Comparator)
  Interventions: Other: Aligners cleansing with Polident Antibacterial Denture Cleaner
- Invisalign Cleaning Crystals® (Active Comparator)
  Interventions: Other: Aligners cleansing with Invisalign Cleaning Crystals
- Geldis® (Active Comparator)
  Interventions: Other: Aligners cleansing with Geldis

INTERVENTIONS:
Other: Aligners cleansing with water — The product is masked in a spraying bottle without any labels. Once a day, for 14 days, the patient sprays the product on the aligner before cleaning it with a soft bristle toothbrush for 1 minute. Afterward, the aligner is rinsed under fresh running water.
  Arms: Water
Other: Aligners cleansing with dish soap Svelto — the product is masked in a transparent bottle without any labels. Once a day, for 14 days, the patient puts the product on the aligner before cleaning it with a soft bristle toothbrush for 1 minute. Afterward, the aligner is rinsed under fresh running water.
  Arms: Dish soap
Other: Aligners cleansing with Polident Antibacterial Denture Cleaner — the product is masked by deleting all labels on the packaging with a black permanent marker. Once a day, for 14 days, the patient dissolves the tablet in a glass full of warm water (30-35 °C), then the aligner is placed inside it for 5 minutes. Afterward the aligner is rinsed under fresh running water.
  Arms: Polident Antibacterial Denture Cleaner®
Other: Aligners cleansing with Invisalign Cleaning Crystals — the product is masked by deleting all labels on the packaging with a black permanent marker. Once a day, for 14 days, the patient dissolves the crystals in a glass full of warm water (30-35 °C) mixing with a spoon for 20 seconds; then, the aligner is placed inside the glass for 15 minutes. Afterward, the aligner is rinsed under fresh running water.
  Arms: Invisalign Cleaning Crystals®
Other: Aligners cleansing with Geldis — the product is masked by deleting all labels on the packaging with a black permanent marker. Once a day, for 14 days, the patient puts the product on the aligner before cleaning it with a soft toothbrush for 1 minute. Afterward, the aligner is rinsed under fresh running water.
  Arms: Geldis®

SUMMARY:
The aim of the study is to evaluate the most efficient product for the cleaning of Invisalign® clear aligners (Align Technology Inc., San Jose, CA, USA) through objective and subjective assessments after the use of 5 different products. For each aligner, one product is used for 2 weeks until all of them are used, therefore 5 different aligners are required for the study. A periodontal evaluation is conducted to assess variations during the time frame of the study.

DETAILED DESCRIPTION:
This randomized clinical trial aims to evaluate the efficacy of 5 different products for the cleansing of Invisalign® clear aligners among the followings:

1. drinking water;
2. dish soap Svelto (Unilever Italia Mkt operations S.r.l.; Roma, IT);
3. Polident Antibacterial Denture Cleaner (GlaxoSmithKline; Philadelphia, Pa, USA);
4. Cleaning Crystals Invisalign® (Align Technology, Inc.; San Jose, CA, USA);
5. Geldis (Kalipharm S.r.l., Alba, IT).

Patients that will sign the informed consent will be enrolled for the study; parents will sign the consent for underage patients.

2 week before the beginning of the orthodontic treatment with Invisalign clear aligners, a professional manual and mechanical removal of supragingival and subgingival deposits of both arches will be performed. At the baseline (T0), the first aligner will be delivered to the patient, that must wear it for 22/24 h except for meals and oral hygiene procedures. One of the 5 cleaning product will be randomly assigned to the patient and toothbrush with silicone bristles (Kalipharm S.r.l., Alba, IT) will be given the cleaning procedures. Patients will be asked to fill in a questionnaire for the subjective appreciation on the cleaning material: the questionnaire presents 19 items evaluating organoleptic and visual characteristics of the aligners and the ease of use of the cleaning method after the first use, after 1 and after 2 weeks. After 2 weeks (T1), patient will be visited again: the questionnaire will be collected, together with the aligner, and a periodontal evaluation on the Ramfjiord teeth will be performed using the following indices: Plaque Index (PI), Bleeding on Probing (BoP), Probing Pocket Depth (PPD), (Gingival Index), BEWE (Basic Erosive Wear Examination), Schiff Air Index. After that, another questionnaire and the following aligner will be given to the patient, another cleaning product will be randomly assigned and another toothbrush will be given. The procedure will be repeated for the following 2 (T2), 4 (T3), 6 (T4) and 8 weeks (T5) until all the cleaning products are tested. All the products will be masked.

JASCO V-750 spectrophotometer (Jasco Corporation, Tokyo, Japan) will be used to evaluate adsorbance for each aligner after the application of the cleaning products. A control value will be calculated using a new clean aligner. The spectrophotometer calculates reflectance values that will be converted in adsorbance values.

Sample size

Sample size was calculated with the following assumptions: ability to detect a clinically relevant difference of 0.0265 in the adsorbance of the clear aligner (primary outcome) of the five groups with an alfa = 0.05 and power = 80%. The assumptions were based on findings of a previous study, with an expected value of 0.190 and a standard deviation of 0.03 for the first group after 2 weeks. Therefore, 20 aligners per each cleaning method were required for the study.

Statistical analysis Statistical analysis will be conducted with R software (R version 3.1.3, R Development Core Team, R Foundation for Statistical Computing, Wien, Austria).

For each variable, Significance for all statistical tests will be predetermined at P<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing orthodontic treatment with Invisalign® clear aligners.

Exclusion Criteria:

* Failing to follow cleaning method instructions
* Failing to fill in the questionnaires

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-07-28 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Change in adsorbance (A) value | Baseline (T0) and after 14 days from baseline (T1)
  The changes in adsorbance values evaluated with a spectrophotometer.
Changes in patient's perception | Baseline (T0) and after 14 days from baseline (T1)
  Through a questionnaire, a subjective evaluation is carried out as regards:
  * the patient's perception of the ease of use of the five products;
  * the difference perceived by the patient in terms of subjective changes in color, smell, taste, cleanness and tactile sensation after the first use, after a week and after 2 weeks of the cleaning method.
  For each of the 19 questions, a mark from 0 (worse mark) to 10 (best mark) will be provided.

SECONDARY OUTCOMES:
Changes in Probing Pocket Depth (PPD) values | Baseline (T0) and after 14 days from baseline (T1)
  PPD is evaluated with a periodontal probe on the facial and lingual surfaces of the Ramfjord teeth in three sites: distal, central and mesial.
Changes in Gingival Index (GI) values | Baseline (T0) and after 14 days from baseline (T1)
  Site-specific assessment of the presence or absence of gingival inflammation.
  Scoring criteria:
  * 0: absence of inflammation;
  * 1: mild inflammation;
  * 2: moderate inflammation;
  * 3: severe inflammation.
Changes in Bleeding on probing (BOP) | Baseline (T0) and after 14 days from baseline (T1)
  Site-specific assessment of the presence or absence of gum bleeding after the insertion of the periodontal probe for the detection of PPD, detected on 4 sites (mesial, distal, vestibular, palatal/lingual).
Change in Schiff Air Index - Dental sensitivity test | Baseline (T0) and after 14 days from baseline (T1)
  Scoring criteria:
  * 0: the subject did not respond to air blasting;
  * 1: the subject responded to air blasting;
  * 2: the subject responded to air blasting and requested discontinuation;
  * 3: the subject responded to air blasting, requested discontinuation and considered the stimulus to be painful.
Change of the BEWE Index Basic Erosive Wear Examination | Baseline (T0) and after 14 days from baseline (T1)
  Scoring criteria:
  * 0: no erosive tooth wear;
  * 1: initial loss of surface texture;
  * 2: distinct defect, hard tissue loss < 50% of the surface area;
  * 3: hard tissue loss ≥ 50% of the surface area.
Change in plaque index (PI): | Baseline (T0) and after 14 days from baseline (T1)
  Site specific assessment of the amount of plaque on dental surfaces; it is detected on facial and lingual surfaces of the Ramfjord teeth.
  Scoring criteria:
  * 0: absence of plaque;
  * 1: plaque revealed on probing;
  * 2: visible layer of plaque on the tooth surface;
  * 3: abundant plaque on tooth surface. Results indicate the index as a percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Scribante, DDS, PhD, Principal Investigator — University of Pavia
Locations (1):
- Unit of Orthodontics and Pediatric Dentistry - Section of Dentistry - Department of Clinical, Surgical, Diagnostic and Pediatrics - University of Pavia, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
Data will be available upon motivated request to the Principal Investigator.